CLINICAL TRIAL: NCT05617755
Title: An Open-label Phase 1 Study to Evaluate the Safety and Efficacy of AB-1015 in Patients With Resistant/Refractory Epithelial Ovarian Cancer
Brief Title: AB-1015, an Integrated Circuit T (ICT) Cell Therapy in Patients With Platinum Resistant Epithelial Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arsenal Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-1015-101
Record Dates: First submitted 2022-11-04; First posted 2022-11-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Ovarian Epithelial; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Neoplasms, Glandular and Epithelial; Ovarian Diseases; Genital Neoplasm, Female; Abdominal Neoplasm; Recurrence
Keywords: ovarian cancer; fallopian tube cancer; primary peritoneal cancer; platinum resistant
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Neoplasms, Glandular and Epithelial; Ovarian Diseases; Genital Neoplasms, Female; Abdominal Neoplasms; Recurrence | interventions — Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AB-1015 (Experimental): Patients receive fludarabine and cyclophosphamide intravenously on days -5 to -3. Patients receive a single dose of AB-1015 intravenously on day 0.
  Interventions: Biological: AB-1015

INTERVENTIONS:
Biological: AB-1015 — autologous T cell therapy
  Other Names: Integrated Circuit T (ICT) cells

SUMMARY:
This is a multi-center, open-label phase 1 dose escalation trial that uses a modified 3+3 design to identify a recommended phase 2 dose (RP2D) of AB-1015 cell product. Backfill cohorts will enroll additional subjects at doses deemed to be safe for a total enrollment of up to 12 subjects per each backfill cohort on the protocol.

DETAILED DESCRIPTION:
This study is intended for the patients who have been diagnosed with Epithelial Ovarian Cancer that either came back or did not improve after platinum treatments (platinum resistant). The purpose of this study is to test the safety of using a new treatment called Integrated Circuit T (ICT) cells (AB-1015 cells) in patients with ovarian cancer. This treatment has not been approved by the Food and Drug Administration.

The goal of this study is to calculate the maximum tolerated dose of the AB-1015 cells. T cells are part of the immune system that protect the body from infection and may help fight cancer. The T cells given in this study will come from the patient and will have a genetic circuit/logic gate put in them that makes them able to recognize alkaline phosphatase, germ line/placental (ALPG/P) and mesothelin (MSLN), 2 proteins on the surface of tumor cells. These logic-gated T cells may help the body's immune system identify and kill cancer cells while sparing normal healthy tissues from toxicity.

The AB-1015 cells are given intravenously, after completing 3 rounds of conditioning chemotherapy administered over 3 consecutive days. Conditioning chemotherapy prepares the body to receive the AB-1015 cells. If they continue to meet the eligibility criteria, AB-1015 cells will be given to them 2 days after the last conditioning chemotherapy round. A single infusion of the AB-1015 cells will be given to the subject intravenously.

After completion of study treatment, patients are followed with serial measurements of safety, tolerability and response.

This is a research study to obtain new information that may help people in the future.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent, advanced, platinum resistant ovarian, fallopian tube, and primary peritoneal cancer and must have a histological diagnosis of a high-grade serous histology.
* a) Platinum resistant disease is defined as progression of disease within six months of platinum regimen.
* Doubling of cancer antigen 125 (CA-125) level on 2 successive measurements may be considered as meeting the definition of disease progression
* b) Have received at least 2 lines of prior therapy including a platinum-based regimen if eligible and a poly-ADP ribose polymerase (PARP) inhibitor if BRCA1/2 mutated. No more than 3 lines of prior therapy for the treatment of platinum resistant disease is permitted.
* Adequate organ function as per protocol definitions.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1.
* Evaluable disease (dose escalation cohorts) or measurable disease (backfill cohorts) at time of enrollment as per protocol definitions.
* Negative pregnancy test for women of childbearing potential. Women of non-childbearing potential are those who have been surgically sterilized, have medically confirmed ovarian failure, or have not had menses within the past 12 months.

Exclusion Criteria:

* Cytotoxic chemotherapy within 14 days of time of cell collection.
* Cytotoxic chemotherapy within 14 days of starting of conditioning chemotherapy.
* New York Heart Association functional class II-IV cardiovascular disability
* Clinically significant pericardial effusion
* Pleural or peritoneal effusion that requires drainage for symptom management within 28 days of screening.
* Active autoimmune disease requiring immunosuppressive therapy or uncontrolled with treatment.
* Untreated brain metastasis.
* Subjects unwilling to participate in an extended safety monitoring period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and dose limiting toxicities (DLTs) | Up to 2 years post treatment
  Toxicity grading will be evaluated according to the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events version 5.0 and monitoring of adverse events. Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) events will be graded according to the criteria outlined in the protocol.
Maximal tolerated dose of AB-1015 | Up to 21 days
  Will be determined by a 3x3 dose escalation study

SECONDARY OUTCOMES:
Number of AB-1015 cells | Up to 1 year post treatment
  Number of AB-1015 cells present in patients treatment with AB-1015
Evidence of anti-tumor activity | Up to 2 years post treatment
  Assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Co-expression of ALPG and MSLN targets on tumor cells | Up to 2 years post treatment
  Assessment by immunohistochemistry (or similar method)

CONTACTS AND LOCATIONS:
Overall Officials: Arsenal Biosciences, Study Director — Arsenal Biosciences
Locations (8):
- United States (8):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - U of Colorado Cancer Center - Anschutz Medical Campus, Aurora, Colorado
  - U of Iowa Health Care, Iowa City, Iowa
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - U of Washington - Fred Hutchinson Cancer Center, Seattle, Washington